CLINICAL TRIAL: NCT04599439
Title: CMR Based Prediction of Ventricular Tachycardia Events in Healed Myocardial Infarction (DEVELOP-VT)
Acronym: DEVELOP-VT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Medico Teknon (Other)
Responsible Party: Principal Investigator, Antonio Berruezo, MD, PhD, Head of Arrhythmia Department & Director of Research and Innovation, Centro Medico Teknon
Other Study IDs: DEVELOP-VT
Record Dates: First submitted 2020-10-17; First posted 2020-10-22 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Myocardial Infarction; Myocardial Infarction Old; Arrhythmias, Cardiac; Ventricular Tachycardia; Ventricular Arrythmia; Sudden Cardiac Death; Sudden Cardiac Death Due to Cardiac Arrhythmia
Keywords: myocardial infarction; cardiac magnetic resonance imaging; scar arrhythmogenicity; ventricular arrhythmias; sudden cardiac death; border zone channels
MeSH Terms: conditions — Myocardial Infarction; Arrhythmias, Cardiac; Tachycardia, Ventricular; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High arrhythmia risk: Patients with a cardiac magnetic resonance-derived border zone channel (BZC) mass > 5.15 g will be considered at highest risk for developing ventricular arrhythmias (VA) or sudden cardiac death (SCD).
  Interventions: Diagnostic Test: Cardiac magnetic resonance imaging
- Low arrhythmia risk: Patients with a cardiac magnetic resonance-derived border zone channel (BZC) mass < 5.15 g will be considered at lowest risk for developing ventricular arrhythmias (VA) or sudden cardiac death (SCD).
  Interventions: Diagnostic Test: Cardiac magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Cardiac magnetic resonance imaging — All patients will undergo a cardiac magnetic resonance test to calculate their border zone channel (BZC) mass. This will not be used to decide further interventions, but all the patients will be treated according to standards of care.

SUMMARY:
Fibrotic tissue is known to be the substrate for the appearance of scar-related reentrant ventricular arrhythmias (VA) in chronic ischemic cardiomyopathy (ICM). Late gadolinium enhancement cardiac magnetic resonance (LGE-CMR) has proven to be a useful technique in the non-invasive characterization of the scarred tissue and the underlying arrhythmogenic substrate. Previous studies identified the presence of significant scarring (> 5% of the left ventricular -LV- mass) is an independent predictor of adverse outcome (all-cause mortality or appropriate ICD discharge for ventricular tachycardia or fibrillation) in patients being considered for implantable cardioverter-defibrillator (ICD) placement. Parallelly, the presence of heterogeneous tissue channels, which correlate with voltage channels after endocardial voltage mapping of the scar, can be more frequently observed in patients suffering from sustained monomorphic ventricular tachycardias (SMVT) than in matched controls for age, sex, infarct location, and left ventricular ejection fraction (LVEF). However, the lack of solid evidence and randomized trials make LVEF still the main decision parameter when assessing suitability for ICD implantation in primary prevention of sudden cardiac death (SCD). In a recent, case-control study, we identified the border zone channel (BZC) mass as the only independent predictor for VT occurrence, after matching for age, sex, LVEF and total scar mass. This BZC mass can be automatically calculated using a commercially available, post-processing imaging platform named ADAS 3D LV (ADAS3D Medical, Barcelona, Spain), with FDA 510(k) Clearance and European Community Mark approval. Thus, CMR-derived BZC mass might be used as an automatically reproducible criterium to reclassify those patients with chronic ICM at highest risk for developing VA/SCD in a relatively short period of approx. 2 years.

In the present cohort study, we sought to evaluate the usefulness of the BZC mass measurement to predict the occurrence of VT events in a prospective, multicenter, unselected series of consecutive chronic ischemic patients without previous arrhythmia evidence, irrespectively of their LVEF.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Chronic (> 3 months after the index coronary event), stable ischemic heart disease, irrespectively of the LVEF.
* Life expectancy of > 1 year with a good functional status.
* Signed informed consent.

Exclusion Criteria:

* Age < 18 years.
* Pregnancy.
* Life expectancy of < 1 year, or bad functional status (NYHA IV functional class).
* Other concomitant structural heart diseases (e.g. congenital, non-ischemic, etc.)
* Previously documented sustained ventricular arrhythmias.
* Impossibility or contraindications to undergo a contrast-enhanced CMR study.
* Concomitant investigation treatments.
* Medical, geographical and social factors that make study participation impractical, and inability to give written informed consent. Patient's refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with chronic (> 3 months after the index coronary event), stable ischemic heart disease, irrespectively of the LVEF, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Ventricular arrhythmias or sudden cardiac death | 2 years
  Clinical composite of cardiac death or any sustained ventricular arrhythmia after a 2-year follow-up period.

SECONDARY OUTCOMES:
Non-cardiac causes of mortality | 2 years
  Death due to non-cardiac conditions
Heart failure hospitalization rate | 2 years
  Hospitalization due to decompensated heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Berruezo, MD, PhD, Principal Investigator — Centro Médico Teknon
Locations (1):
- Antonio Berruezo, MD, PhD, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Bakker JM, van Capelle FJ, Janse MJ, Wilde AA, Coronel R, Becker AE, Dingemans KP, van Hemel NM, Hauer RN. Reentry as a cause of ventricular tachycardia in patients with chronic ischemic heart disease: electrophysiologic and anatomic correlation. Circulation. 1988 Mar;77(3):589-606. doi: 10.1161/01.cir.77.3.589. PMID 3342490
- [Background] Wu E, Judd RM, Vargas JD, Klocke FJ, Bonow RO, Kim RJ. Visualisation of presence, location, and transmural extent of healed Q-wave and non-Q-wave myocardial infarction. Lancet. 2001 Jan 6;357(9249):21-8. doi: 10.1016/S0140-6736(00)03567-4. PMID 11197356
- [Background] Schmidt A, Azevedo CF, Cheng A, Gupta SN, Bluemke DA, Foo TK, Gerstenblith G, Weiss RG, Marban E, Tomaselli GF, Lima JA, Wu KC. Infarct tissue heterogeneity by magnetic resonance imaging identifies enhanced cardiac arrhythmia susceptibility in patients with left ventricular dysfunction. Circulation. 2007 Apr 17;115(15):2006-14. doi: 10.1161/CIRCULATIONAHA.106.653568. Epub 2007 Mar 26. PMID 17389270
- [Background] Yan AT, Shayne AJ, Brown KA, Gupta SN, Chan CW, Luu TM, Di Carli MF, Reynolds HG, Stevenson WG, Kwong RY. Characterization of the peri-infarct zone by contrast-enhanced cardiac magnetic resonance imaging is a powerful predictor of post-myocardial infarction mortality. Circulation. 2006 Jul 4;114(1):32-9. doi: 10.1161/CIRCULATIONAHA.106.613414. Epub 2006 Jun 26. PMID 16801462
- [Background] Klem I, Weinsaft JW, Bahnson TD, Hegland D, Kim HW, Hayes B, Parker MA, Judd RM, Kim RJ. Assessment of myocardial scarring improves risk stratification in patients evaluated for cardiac defibrillator implantation. J Am Coll Cardiol. 2012 Jul 31;60(5):408-20. doi: 10.1016/j.jacc.2012.02.070. PMID 22835669
- [Background] Perez-David E, Arenal A, Rubio-Guivernau JL, del Castillo R, Atea L, Arbelo E, Caballero E, Celorrio V, Datino T, Gonzalez-Torrecilla E, Atienza F, Ledesma-Carbayo MJ, Bermejo J, Medina A, Fernandez-Aviles F. Noninvasive identification of ventricular tachycardia-related conducting channels using contrast-enhanced magnetic resonance imaging in patients with chronic myocardial infarction: comparison of signal intensity scar mapping and endocardial voltage mapping. J Am Coll Cardiol. 2011 Jan 11;57(2):184-94. doi: 10.1016/j.jacc.2010.07.043. PMID 21211689
- [Background] Moss AJ, Zareba W, Hall WJ, Klein H, Wilber DJ, Cannom DS, Daubert JP, Higgins SL, Brown MW, Andrews ML; Multicenter Automatic Defibrillator Implantation Trial II Investigators. Prophylactic implantation of a defibrillator in patients with myocardial infarction and reduced ejection fraction. N Engl J Med. 2002 Mar 21;346(12):877-83. doi: 10.1056/NEJMoa013474. Epub 2002 Mar 19. PMID 11907286
- [Background] Bardy GH, Lee KL, Mark DB, Poole JE, Packer DL, Boineau R, Domanski M, Troutman C, Anderson J, Johnson G, McNulty SE, Clapp-Channing N, Davidson-Ray LD, Fraulo ES, Fishbein DP, Luceri RM, Ip JH; Sudden Cardiac Death in Heart Failure Trial (SCD-HeFT) Investigators. Amiodarone or an implantable cardioverter-defibrillator for congestive heart failure. N Engl J Med. 2005 Jan 20;352(3):225-37. doi: 10.1056/NEJMoa043399. PMID 15659722
- [Background] Andreu D, Ortiz-Perez JT, Fernandez-Armenta J, Guiu E, Acosta J, Prat-Gonzalez S, De Caralt TM, Perea RJ, Garrido C, Mont L, Brugada J, Berruezo A. 3D delayed-enhanced magnetic resonance sequences improve conducting channel delineation prior to ventricular tachycardia ablation. Europace. 2015 Jun;17(6):938-45. doi: 10.1093/europace/euu310. Epub 2015 Jan 23. PMID 25616406
- [Background] Andreu D, Berruezo A, Ortiz-Perez JT, Silva E, Mont L, Borras R, de Caralt TM, Perea RJ, Fernandez-Armenta J, Zeljko H, Brugada J. Integration of 3D electroanatomic maps and magnetic resonance scar characterization into the navigation system to guide ventricular tachycardia ablation. Circ Arrhythm Electrophysiol. 2011 Oct;4(5):674-83. doi: 10.1161/CIRCEP.111.961946. Epub 2011 Aug 31. PMID 21880674
- [Background] Zeitler EP, Al-Khatib SM, Friedman DJ, Han JY, Poole JE, Bardy GH, Bigger JT, Buxton AE, Moss AJ, Lee KL, Dorian P, Cappato R, Kadish AH, Kudenchuk PJ, Mark DB, Inoue LYT, Sanders GD. Predicting appropriate shocks in patients with heart failure: Patient level meta-analysis from SCD-HeFT and MADIT II. J Cardiovasc Electrophysiol. 2017 Nov;28(11):1345-1351. doi: 10.1111/jce.13307. Epub 2017 Aug 23. PMID 28744959
- [Background] Acosta J, Fernandez-Armenta J, Borras R, Anguera I, Bisbal F, Marti-Almor J, Tolosana JM, Penela D, Andreu D, Soto-Iglesias D, Evertz R, Matiello M, Alonso C, Villuendas R, de Caralt TM, Perea RJ, Ortiz JT, Bosch X, Serra L, Planes X, Greiser A, Ekinci O, Lasalvia L, Mont L, Berruezo A. Scar Characterization to Predict Life-Threatening Arrhythmic Events and Sudden Cardiac Death in Patients With Cardiac Resynchronization Therapy: The GAUDI-CRT Study. JACC Cardiovasc Imaging. 2018 Apr;11(4):561-572. doi: 10.1016/j.jcmg.2017.04.021. Epub 2017 Aug 2. PMID 28780194
- [Background] Ikeda T, Yoshino H, Sugi K, Tanno K, Shimizu H, Watanabe J, Kasamaki Y, Yoshida A, Kato T. Predictive value of microvolt T-wave alternans for sudden cardiac death in patients with preserved cardiac function after acute myocardial infarction: results of a collaborative cohort study. J Am Coll Cardiol. 2006 Dec 5;48(11):2268-74. doi: 10.1016/j.jacc.2006.06.075. Epub 2006 Nov 9. PMID 17161258
- [Background] Gatzoulis KA, Tsiachris D, Arsenos P, Antoniou CK, Dilaveris P, Sideris S, Kanoupakis E, Simantirakis E, Korantzopoulos P, Goudevenos I, Flevari P, Iliodromitis E, Sideris A, Vassilikos V, Fragakis N, Trachanas K, Vernardos M, Konstantinou I, Tsimos K, Xenogiannis I, Vlachos K, Saplaouras A, Triantafyllou K, Kallikazaros I, Tousoulis D. Arrhythmic risk stratification in post-myocardial infarction patients with preserved ejection fraction: the PRESERVE EF study. Eur Heart J. 2019 Sep 14;40(35):2940-2949. doi: 10.1093/eurheartj/ehz260. PMID 31049557